CLINICAL TRIAL: NCT00025272
Title: Phase II Study of Sequential Topotecan-Carboplatin-Etoposide in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: REBACDR0000068945; CCCWFU-62300; NCI-5333
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Etoposide; Topotecan; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: etoposide
Drug: topotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining topotecan, carboplatin, and etoposide in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity profile and maximum tolerated dose of sequential topotecan, carboplatin, and etoposide in patients with chemotherapy-naive extensive stage small cell lung cancer. (Phase I closed to accrual as of 04/04/2003).
* Determine the response rate and duration of response in patients with treated with this regimen.
* Determine the failure-free and overall survival of patients treated with this regimen.
* Determine the pharmacokinetics and pharmacodynamics of topotecan and etoposide on this schedule in these patients.

OUTLINE: This is a dose-escalation, multicenter study of topotecan and etoposide. (Phase I closed to accrual as of 04/04/2003).

Patients receive oral topotecan on days 1-5, carboplatin IV over 30 minutes on day 6, and oral etoposide on days 6-10. Treatment continues every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) or partial response after the second course receive up to 4 additional courses. Patients with brain metastases at initial presentation undergo whole-brain irradiation before the chemotherapy regimen. Patients without brain metastases at initial presentation who achieve CR undergo prophylactic whole-brain irradiation.

Sequential dose escalation of topotecan is followed by sequential dose escalation of etoposide. Cohorts of 3-6 patients receive escalating doses of topotecan and then etoposide until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. (Phase I closed to accrual as of 04/04/2003). In the phase II part of study, an additional 11-40 patients are accrued to receive topotecan, carboplatin, and etoposide at the MTD.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A maximum of 50 patients (3-10 for phase I and 11-40 for phase II) will be accrued for this study. (Phase I closed to accrual as of 04/04/2003)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed extensive stage small cell lung cancer
* Measurable or evaluable disease

  * Pleural effusions allowed, but not considered measurable or evaluable disease
* Brain metastases allowed provided neurologically stable at study entry

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow capsules
* No concurrent or prior malignancy within the past 5 years except inactive nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No other serious medical or psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy for brain metastasis allowed
* No other prior radiotherapy
* No other concurrent radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-11-01 (Actual); Primary Completion 2005-01-18 (Actual); Study Completion 2005-01-18 (Actual)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Duration of response
Failure-free and overall survival
Pharmacokinetics and pharmacodynamics of topotecan and etoposide

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (5):
- United States (5):
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - MBCCOP - Massey Cancer Center, Richmond, Virginia